CLINICAL TRIAL: NCT03913299
Title: Frailty Assessment by Edmonton Frail Scale to Predict Outcome in Patients Undergoing Cardiovascular Surgery "Frail Heart" Study.
Brief Title: Frailty Assessment by Edmonton Frail Scale to Predict Outcome in Patients Undergoing Cardiovascular Surgery
Acronym: FRAIL-HEART
Status: Active, not recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Frail Heart; 2019/26FEV/094 (Other: CEHF)
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Frail Elderly Syndrome; Frailty; Surgery
Keywords: Frailty; Cardiac surgery; Vascular surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess frailty of patients admited for cardio-vascular surgery in Cliniques Universitaires Saint Luc in Brussels. And analyse the correlation between frailty, functionnal decline and postoperative mortality.

DETAILED DESCRIPTION:
Frailty is a state of loss of functional reserve resulting in an increased vulnerability to a stressor event. From a pathophysiological point of view, it is an accelerated decrease in physiological reserve related to ageing.

Currently, evaluation of the outcome after cardiac surgery is commonly based on scores not taking into account the concept of frailty (Society of Thoracic Surgeons (STS) and Eurosore II) Recent studies have shown an independent association between post cardiac surgery mortality and pre-operative frailty. Beyond cardiac surgery, frailty has been shown to be associated with higher mortality and morbidity among intensive care unit (ICU) patients. Frailty is commonly assessed for patients older than 75 years of age but the prevalence in younger patients admitted to the hospital is significant. There is therefore need to evaluate all patients for frailty in the preoperative period.

Since the Edmonton Frail Scale (EFS) allows easy screening of all frailty domains, we hypothesized that it could be a reliable and feasible score to assess preoperative frailty and to predict postoperative morbidity and mortality.

Objectives:

The primary objective of this study is to evaluate preoperative frailty in all adult patients undergoing cardiac and vascular surgery.

The secondary objectives are:

* to evaluate the association between frailty and postoperative mortality.
* to evaluate the association between frailty and postoperative functional decline (nursing home admission or care dependency)
* to evaluate impact of each frailty domain on the post-operative outcomes (mortality and functional decline)
* to evaluate how to integrate frailty with the others preoperative clinical parameters to better predict postoperative outcome

Measurement:

Assessment of frailty will be performed using EFS. Other clinical conditions related to frailty will be collected: Body Mass Idex (BMI), tobacco use, alcohol consumption, preoperative albumin and pre-albumin level. STS and Eurosore II will be systematically calculated.

A one-year follow-up will assess the following parameters:

* all-cause mortality
* functional decline with admission to a nursing home or care dependency. Care dependency will be defined by a Katz index more than 0 [19].

Follow-up will be realized by a phone call to the patient, his relatives or his general practitioner.

Based on a prevalence of frailty of 11%, we have determined that the enrollment of a minimum of 2080 patients would provide a power of 80% at a significance level of 5% to detect a difference of 5% mortality at one year between frail and non-frail patients.

ELIGIBILITY:
Inclusion Criteria:

* Any cardiac surgery under cardiopulmonary bypass
* Any vascular surgery

Exclusion Criteria:

* Salvage surgery
* Cirrhosis CHILD B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients older than 18 years of age admitted for cardiac surgery or vascular surgery in Cliniques Universitaires Saint-Luc in Brussels will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2080 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
Functionnal decline | 1 year
  Admission to a nursing home (yes or no) or care dependency (defined by a Katz index higher than 0/6)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Dechamps, MD, Principal Investigator — St Luc University Hospital UCLouvain
Locations (3):
- Belgium (3):
  - St Luc University Hospital UCLouvain, Brussels
  - Grand Hopital Charleroi, Charleroi
  - Centre Hospitalier Universitaire de Liège, Liège

REFERENCES:
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Nashef SA, Roques F, Sharples LD, Nilsson J, Smith C, Goldstone AR, Lockowandt U. EuroSCORE II. Eur J Cardiothorac Surg. 2012 Apr;41(4):734-44; discussion 744-5. doi: 10.1093/ejcts/ezs043. Epub 2012 Feb 29. PMID 22378855
- [Background] Anderson RP. First publications from the Society of Thoracic Surgeons National Database. Ann Thorac Surg. 1994 Jan;57(1):6-7. doi: 10.1016/0003-4975(94)90355-7. No abstract available. PMID 8279920
- [Background] Sundermann S, Dademasch A, Praetorius J, Kempfert J, Dewey T, Falk V, Mohr FW, Walther T. Comprehensive assessment of frailty for elderly high-risk patients undergoing cardiac surgery. Eur J Cardiothorac Surg. 2011 Jan;39(1):33-7. doi: 10.1016/j.ejcts.2010.04.013. PMID 20627611
- [Background] Bagshaw SM, Stelfox HT, Johnson JA, McDermid RC, Rolfson DB, Tsuyuki RT, Ibrahim Q, Majumdar SR. Long-term association between frailty and health-related quality of life among survivors of critical illness: a prospective multicenter cohort study. Crit Care Med. 2015 May;43(5):973-82. doi: 10.1097/CCM.0000000000000860. PMID 25668751
- [Background] Ferrante LE, Pisani MA, Murphy TE, Gahbauer EA, Leo-Summers LS, Gill TM. The Association of Frailty With Post-ICU Disability, Nursing Home Admission, and Mortality: A Longitudinal Study. Chest. 2018 Jun;153(6):1378-1386. doi: 10.1016/j.chest.2018.03.007. Epub 2018 Mar 17. PMID 29559308
- [Background] Le Maguet P, Roquilly A, Lasocki S, Asehnoune K, Carise E, Saint Martin M, Mimoz O, Le Gac G, Somme D, Cattenoz C, Feuillet F, Malledant Y, Seguin P. Prevalence and impact of frailty on mortality in elderly ICU patients: a prospective, multicenter, observational study. Intensive Care Med. 2014 May;40(5):674-82. doi: 10.1007/s00134-014-3253-4. Epub 2014 Mar 21. PMID 24651884
- [Background] Muscedere J, Waters B, Varambally A, Bagshaw SM, Boyd JG, Maslove D, Sibley S, Rockwood K. The impact of frailty on intensive care unit outcomes: a systematic review and meta-analysis. Intensive Care Med. 2017 Aug;43(8):1105-1122. doi: 10.1007/s00134-017-4867-0. Epub 2017 Jul 4. PMID 28676896
- [Background] Smart R, Carter B, McGovern J, Luckman S, Connelly A, Hewitt J, Quasim T, Moug S. Frailty Exists in Younger Adults Admitted as Surgical Emergency Leading to Adverse Outcomes. J Frailty Aging. 2017;6(4):219-223. doi: 10.14283/jfa.2017.28. PMID 29165541
- [Background] Bagshaw M, Majumdar SR, Rolfson DB, Ibrahim Q, McDermid RC, Stelfox HT. A prospective multicenter cohort study of frailty in younger critically ill patients. Crit Care. 2016 Jun 6;20(1):175. doi: 10.1186/s13054-016-1338-x. PMID 27263535
- [Background] Brummel NE, Bell SP, Girard TD, Pandharipande PP, Jackson JC, Morandi A, Thompson JL, Chandrasekhar R, Bernard GR, Dittus RS, Gill TM, Ely EW. Frailty and Subsequent Disability and Mortality among Patients with Critical Illness. Am J Respir Crit Care Med. 2017 Jul 1;196(1):64-72. doi: 10.1164/rccm.201605-0939OC. PMID 27922747
- [Background] Sundermann S, Dademasch A, Rastan A, Praetorius J, Rodriguez H, Walther T, Mohr FW, Falk V. One-year follow-up of patients undergoing elective cardiac surgery assessed with the Comprehensive Assessment of Frailty test and its simplified form. Interact Cardiovasc Thorac Surg. 2011 Aug;13(2):119-23; discussion 123. doi: 10.1510/icvts.2010.251884. Epub 2011 Mar 4. PMID 21378017
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Rolfson DB, Majumdar SR, Tsuyuki RT, Tahir A, Rockwood K. Validity and reliability of the Edmonton Frail Scale. Age Ageing. 2006 Sep;35(5):526-9. doi: 10.1093/ageing/afl041. Epub 2006 Jun 6. No abstract available. PMID 16757522
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] Kobe AR, Meyer A, Elmubarak H, Kempfert J, Pavicevic J, Maisano F, Walther T, Falk V, Sundermann SH. Frailty Assessed by the FORECAST Is a Valid Tool to Predict Short-Term Outcome After Transcatheter Aortic Valve Replacement. Innovations (Phila). 2016 Nov/Dec;11(6):407-413. doi: 10.1097/IMI.0000000000000321. PMID 27926626
- [Background] Reichart D, Rosato S, Nammas W, Onorati F, Dalen M, Castro L, Gherli R, Gatti G, Franzese I, Faggian G, De Feo M, Khodabandeh S, Santarpino G, Rubino AS, Maselli D, Nardella S, Salsano A, Nicolini F, Zanobini M, Saccocci M, Bounader K, Kinnunen EM, Tauriainen T, Airaksinen J, Seccareccia F, Mariscalco G, Ruggieri VG, Perrotti A, Biancari F. Clinical frailty scale and outcome after coronary artery bypass grafting. Eur J Cardiothorac Surg. 2018 Dec 1;54(6):1102-1109. doi: 10.1093/ejcts/ezy222. PMID 29897529